CLINICAL TRIAL: NCT07404124
Title: Comparison of Sensory and Motor Block Characteristics and Postoperative Analgesic Consumption After Ultrasound-Guided Ankle Block in Diabetic and Non-Diabetic Patients Undergoing Lower Extremity Surgery
Brief Title: Effects of Ankle Block on Postoperative Analgesia in Diabetic and Non-Diabetic Patients
Acronym: ANKLE-DM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, dogameric, MD, Anesthesiology Specialist, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FSM-SUAM-ANKLEBLOCK-2026
Record Dates: First submitted 2026-01-29; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus; Diabetic Neuropathy; Postoperative Pain Management
Keywords: Ankle Block; Ultrasound-Guided Regional Anesthesia; Peripheral Nerve Block; Diabetes Mellitus; Diabetic Neuropathy; Glycemic Control; Postoperative Analgesia; HBA1C; Lower Extremity Surgery; Opioid Consumption
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective observational study with no intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational Cohort (Experimental): Adult patients undergoing lower extremity surgery under routine ultrasound-guided ankle block as part of standard clinical care. Participants are not assigned to any intervention for research purposes.
  Interventions: Procedure: Ultrasound-Guided Ankle Block

INTERVENTIONS:
Procedure: Ultrasound-Guided Ankle Block — Ultrasound-guided ankle block performed as part of routine clinical practice for anesthesia and postoperative analgesia. The procedure is not administered as an experimental intervention and is not assigned by the study protocol

SUMMARY:
This prospective observational study aims to evaluate the effects of ultrasound-guided ankle block on sensory and motor block characteristics and postoperative analgesic outcomes in patients undergoing lower extremity surgery. The study will compare diabetic and non-diabetic patients and will also assess the impact of glycemic control on block onset time and postoperative analgesic consumption.

Ankle block is commonly used in patients undergoing foot and ankle surgery, particularly in those with diabetes, peripheral neuropathy, or vascular disease, when general or neuraxial anesthesia may not be suitable. Previous studies suggest that diabetic neuropathy and impaired glycemic control may influence the onset and duration of peripheral nerve blocks.

Adult patients scheduled for lower extremity surgery under ankle block will be included. All procedures will be performed as part of routine clinical care, and no additional interventions will be applied for research purposes. Sensory and motor block onset times, postoperative pain scores, opioid consumption within the first 24 hours, and patient and surgeon satisfaction will be recorded.

The results of this study are expected to provide clinically relevant information regarding the effects of diabetes and glycemic control on ankle block characteristics and postoperative analgesia.

DETAILED DESCRIPTION:
Diabetes mellitus is a common chronic metabolic disease, and its increasing prevalence has led to a rise in diabetes-related complications. Diabetic neuropathy is one of the most frequent complications and is associated with structural and functional changes in peripheral nerves, including axonal degeneration and demyelination. These alterations may affect the onset, duration, and quality of peripheral nerve blocks.

Previous clinical and experimental studies have demonstrated that peripheral nerve blocks in patients with diabetic neuropathy may have longer duration and altered onset times compared to non-diabetic patients. Proposed mechanisms include changes in sodium and potassium channel function, delayed clearance of local anesthetics, and reduced microvascular absorption due to diabetic microangiopathy.

Ultrasound-guided ankle block is a commonly used regional anesthesia technique for foot and ankle surgeries, particularly in patients with diabetic foot ulcers, wound debridement, or minor amputations. It provides effective anesthesia and postoperative analgesia while avoiding the potential risks of general or neuraxial anesthesia in high-risk patients.

This study is designed as a single-center, prospective, observational study conducted at Fatih Sultan Mehmet Training and Research Hospital. Adult patients scheduled for lower extremity surgery under ultrasound-guided ankle block between January 2026 and October 2026 will be included after obtaining written informed consent. No additional interventions beyond routine clinical practice will be performed.

The ankle block will be administered preoperatively under ultrasound guidance by an experienced anesthesiologist using a standardized local anesthetic mixture. Sensory and motor block assessments will be performed using pinprick testing and motor function evaluation. Block onset times and block resolution times will be recorded.

Postoperative outcomes will include pain scores assessed using the Visual Analog Scale (VAS), total opioid consumption within the first 24 hours (expressed as morphine equivalents), time to first analgesic request, and the need for rescue analgesia. Patient and surgeon satisfaction will be evaluated using a 10-point numerical rating scale.

Patients will be categorized based on diabetes status and further subgrouped according to glycemic control using HbA1c levels (<7.5% and ≥7.5%). Outcomes will be compared between diabetic and non-diabetic patients and between glycemic control subgroups to evaluate the effect of diabetes and metabolic control on ankle block characteristics and postoperative analgesic outcomes.

The findings of this study are expected to contribute to a better understanding of regional anesthesia outcomes in diabetic patients and may help optimize anesthetic management strategies in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Patients scheduled for lower extremity surgery under ultrasound-guided ankle block as part of routine clinical care.
* Patients able to provide written informed consent.
* Availability of complete perioperative data including blood glucose levels, -HbA1c values, pain scores, and postoperative analgesic consumption.

Exclusion Criteria:

* Refusal or inability to provide informed consent.
* Failure of ankle block requiring conversion to another anesthesia technique.
* Known coagulation disorders contraindicating peripheral nerve block.
* Active infection at the site of block application.
* Chronic opioid or analgesic use, chronic alcohol use, or substance abuse.
* History of diabetic ketoacidosis or hyperosmolar hyperglycemic state.
* Severe renal or hepatic insufficiency.
* Known allergy to local anesthetics such as lidocaine or bupivacaine.
* Inability to perform perioperative blood glucose monitoring.
* Cognitive impairment or psychiatric conditions interfering with study participation or data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Sensory Block Onset Time | From block completion up to 30 minutes after block administration
  Time from completion of ultrasound-guided ankle block to the onset of sensory block, assessed using pinprick testing (score 0: no sensation, 1: reduced sensation, 2: normal sensation).

SECONDARY OUTCOMES:
Motor Block Onset Time | From block completion up to 30 minutes after block administration
  Time from completion of ankle block to onset of motor block, assessed by ankle dorsiflexion and plantarflexion strength, measured in minutes.
Total Opioid Consumption in the First 24 Hours | First 24 hours after surgery
  Total amount of opioid analgesics consumed within the first 24 hours postoperatively, calculated as intravenous morphine equivalents in milligrams.
Postoperative Pain Scores | At 6, 12, and 24 hours after surgery
  Postoperative pain intensity assessed using the Visual Analog Scale (VAS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates worst imaginable pain. Higher scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: doga meric yukselen, MD, Principal Investigator — ISTANBUL PROVINCIAL HEALTH DIRECTORATE FATIH SULTAN MEHMET TRAINING AND RESEARCH HOSPITAL
Locations (1):
- Istanbul Provincial Health Directorate Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)